CLINICAL TRIAL: NCT07257952
Title: An Observational Study on the Risk of Adverse Maternal and Infant Outcomes Associated With Respiratory Viral Infections Before and During Early Pregnancy
Brief Title: APOs Associated With Respiratory Viral Infections Before and During Early Pregnancy
Acronym: APO
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, China (Other)
Responsible Party: Principal Investigator, Mei Kang, Associate Professor, Shanghai General Hospital, China
Other Study IDs: 2025-K434
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Viral Infections; Adverse Pregnancy Outcomes
Keywords: Adverse pregnancy outcome; Preterm birth; Gestational diabetes mullitus; Respiratory Viral Infection
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Respiratory viral infections cohort: Women with respiratory viral infections during 6 months before pregnancy or early pregnancy
- Control cohort: Women without respiratory viral infections during 6 months before pregnancy or early pregnancy

SUMMARY:
Adverse pregnancy outcomes (APOs) are a collection of conditions that have short-term and long-term effects of complications related to pregnancy and childbirth on pregnant women and their fetuses, including hypertensive disorders of pregnancy, gestational diabetes, preterm birth, large for gestational age, among others. Nearly 30% of all women experience an adverse pregnancy outcome during their reproductive years. Although, respiratory viral infections with epidemic and pandemic potential pose an omnipresent threat to public health, research focusing specifically on the maternal-infant population remains relatively scarce.

Studies conducted in USA found that among pregnant women infected with influenza, the proportion of those with gestational hypertension or diabetes was higher than in pregnant women without influenza infection (13.9% vs. 11.1%).

Research on the impact of respiratory viral infections on perinatal outcomes in China is limited, and we aim to establish of a large-scale, retroprospective maternal-child cohorts. This cohort study will systematically collect longitudinal data (e.g., detailed clinical history, timing of infection/vaccination, complication of pregnancy, and APOs) to assess the risk of respiratory viral infections to APOs, as well as facilitate multidisciplinary research.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Age 20 to 45 years old;
* Physician-diagnosed acute respiratory viral infection occurring within 6 months before pregnancy and/or at <24 weeks of gestation.

Exclusion Criteria:

* Pregestational T1D or T2D;
* Long-term use of immunosuppressants or glucocorticoids;
* Diseases that severely affect immune or metabolic function (e.g., HIV, SLE, rheumatoid arthritis);
* Severe mental illness or cognitive impairment;
* Women whose electronic medical records lack GDM screening and delivery records.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women who are planning to conceive or pregnant women.
Study Population: Women who are planning to conceive or pregnant women.
Sampling Method: Non-Probability Sample
Enrollment: 1440 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
incidence of gestational diabetes mallitus | 28 weeks of gestation
  incidence of gestational diabetes mallitus according to International Association of Diabetes and Pregnancy Study Groups consensus if any one of the plasma glucose values is met or exceeded during a 75g oral glucose tolerance test (OGTT) at 20 to 28 gestational weeks.

SECONDARY OUTCOMES:
incidence of preterm birth | 37 gestational weeks
  incidence of any births that occur before 37 completed weeks of gestation

IPD SHARING:
Plan to Share IPD: No
IPD can be requested by sending an email to the corresponding author.

REFERENCES:
- [Background] Liong S, Oseghale O, To EE, Brassington K, Erlich JR, Luong R, Liong F, Brooks R, Martin C, O'Toole S, Vinh A, O'Neill LAJ, Bozinovski S, Vlahos R, Papagianis PC, O'Leary JJ, Brooks DA, Selemidis S. Influenza A virus causes maternal and fetal pathology via innate and adaptive vascular inflammation in mice. Proc Natl Acad Sci U S A. 2020 Oct 6;117(40):24964-24973. doi: 10.1073/pnas.2006905117. Epub 2020 Sep 21. PMID 32958663
- [Background] Gonzalez-Ricon RJ, Otero AM, Chalen I, Savas JN, Adetunji S, Antonson AM. Influenza A virus infection during pregnancy increases transfer of maternal bloodborne molecules to fetal tissues. Brain Behav Immun. 2025 Nov;130:106069. doi: 10.1016/j.bbi.2025.106069. Epub 2025 Aug 6. PMID 40780523
- [Background] Oseghale O, Liong S, Coward-Smith M, To EE, Erlich JR, Luong R, Liong F, Miles M, Norouzi S, Martin C, O'Toole S, Brooks RD, Bozinovski S, Vlahos R, O'Leary JJ, Brooks DA, Selemidis S. Influenza A virus elicits peri-vascular adipose tissue inflammation and vascular dysfunction of the aorta in pregnant mice. PLoS Pathog. 2022 Aug 5;18(8):e1010703. doi: 10.1371/journal.ppat.1010703. eCollection 2022 Aug. PMID 35930608
- [Background] Celik IH, Tanacan A, Canpolat FE. Neonatal outcomes of maternal prenatal coronavirus infection. Pediatr Res. 2024 Jan;95(2):445-455. doi: 10.1038/s41390-023-02950-2. Epub 2023 Dec 6. PMID 38057579
- [Background] Wang J, Liu W, Zhuang Y, Yang J, Zhao Y, Hong A, Du J, Kong H, Wang J, Jiang Y, Wang Y. Influenza A virus infection disrupts the function of syncytiotrophoblast cells and contributes to adverse pregnancy outcomes. J Med Virol. 2024 Jun;96(6):e29687. doi: 10.1002/jmv.29687. PMID 38783821
- [Background] Wang X, Li Y, Shi T, Bont LJ, Chu HY, Zar HJ, Wahi-Singh B, Ma Y, Cong B, Sharland E, Riley RD, Deng J, Figueras-Aloy J, Heikkinen T, Jones MH, Liese JG, Markic J, Mejias A, Nunes MC, Resch B, Satav A, Yeo KT, Simoes EAF, Nair H; Respiratory Virus Global Epidemiology Network; RESCEU investigators. Global disease burden of and risk factors for acute lower respiratory infections caused by respiratory syncytial virus in preterm infants and young children in 2019: a systematic review and meta-analysis of aggregated and individual participant data. Lancet. 2024 Mar 30;403(10433):1241-1253. doi: 10.1016/S0140-6736(24)00138-7. Epub 2024 Feb 14. PMID 38367641
- [Background] Kittikraisak W, Mohanty S, Klungthong C, Macareo L, Rawangban B, Tomyabatra K, Srisantiroj N, Phadungkiatwatana P, Chotpitayasunondh T, Kanjanapattanakul W, Mott JA, Kim L, Dawood FS. Antenatal Respiratory Syncytial Virus and Human Metapneumovirus Illness Rates Among Pregnant Women in Thailand and the Association Between Antenatal Respiratory Syncytial Virus and Perinatal Outcomes: A Prospective Cohort Study. J Infect Dis. 2025 Oct 15;232(4):e651-e655. doi: 10.1093/infdis/jiaf165. PMID 40176473
- [Background] Garcia-Aguilar P, Rolle V, Serrano B, Rodo C, Garcia-Ruiz I, Garcia-Manau P, Farras A, Illan L, Moreno E, Dalmau M, Roldan E, Sirvent E, Temprado J, Seminario N, Fernandez-Hidalgo N, Sulleiro E, Balcells J, Ferrer-Costa R, Maiz N, Carreras E, Suy A, Mendoza M. Effect of SARS-CoV-2 infection on perinatal outcomes by disease severity and trimester of pregnancy: A prospective cohort study. J Gynecol Obstet Hum Reprod. 2026 Jan;55(1):103058. doi: 10.1016/j.jogoh.2025.103058. Epub 2025 Oct 23. PMID 41139067
- [Background] Engjom HM, Ramakrishnan R, Vousden N, Bunch K, Morris E, Simpson N, Gale C, O'Brien P, Quigley M, Brocklehurst P, Kurinczuk JJ, Knight M. Perinatal outcomes after admission with COVID-19 in pregnancy: a UK national cohort study. Nat Commun. 2024 Apr 15;15(1):3234. doi: 10.1038/s41467-024-47181-z. PMID 38622110
- [Background] Zare F, Karimi A, Daliri S. Complications in Pregnant Women and Newborns Before and During the COVID-19 Pandemic. Iran J Nurs Midwifery Res. 2024 Jan 9;29(1):91-97. doi: 10.4103/ijnmr.ijnmr_252_22. eCollection 2024 Jan-Feb. PMID 38333333
- [Background] Sun Y, Luo X, Chen N, Xie L, Hu S, Zhou M, Wang L, Wang L, Li X, Yang Z, Yi P, Xu J. Impact of maternal COVID-19 infection on offspring immunity and maternal-fetal outcomes at different pregnancy stages: a cohort study. BMC Pregnancy Childbirth. 2025 Feb 28;25(1):219. doi: 10.1186/s12884-025-07323-7. PMID 40022096
- [Background] Wang Y, Guo Z, Ye B, Liu L, Mao X, Luo Y, Gao S, He G, Bian S. Association of SARS-CoV-2 Infection during Early Weeks of Gestation with Situs Inversus. N Engl J Med. 2023 Nov 2;389(18):1722-1724. doi: 10.1056/NEJMc2309215. No abstract available. PMID 37913512
- [Background] Conde-Agudelo A, Romero R. SARS-CoV-2 infection during pregnancy and risk of preeclampsia: a systematic review and meta-analysis. Am J Obstet Gynecol. 2022 Jan;226(1):68-89.e3. doi: 10.1016/j.ajog.2021.07.009. Epub 2021 Jul 21. PMID 34302772
- [Background] Camps J, Iftimie S, Jimenez-Franco A, Castro A, Joven J. Metabolic Reprogramming in Respiratory Viral Infections: A Focus on SARS-CoV-2, Influenza, and Respiratory Syncytial Virus. Biomolecules. 2025 Jul 16;15(7):1027. doi: 10.3390/biom15071027. PMID 40723899
- [Background] Darweesh M, Mohammadi S, Rahmati M, Al-Hamadani M, Al-Harrasi A. Metabolic reprogramming in viral infections: the interplay of glucose metabolism and immune responses. Front Immunol. 2025 May 16;16:1578202. doi: 10.3389/fimmu.2025.1578202. eCollection 2025. PMID 40453076
- [Background] Lee H, Yoon D, Kim JH, Noh Y, Joo EJ, Han JY, Choe YJ, Shin JY. Association of Influenza Vaccination During Pregnancy with Health Outcomes in Mothers and Children: A Population-Based Cohort Study. Clin Pharmacol Ther. 2025 May;117(5):1381-1392. doi: 10.1002/cpt.3565. Epub 2025 Jan 23. PMID 39854110
- [Background] Trotta F, Da Cas R, Spila Alegiani S, Gramegna M, Venegoni M, Zocchetti C, Traversa G. Evaluation of safety of A/H1N1 pandemic vaccination during pregnancy: cohort study. BMJ. 2014 May 29;348:g3361. doi: 10.1136/bmj.g3361. PMID 24874845
- [Background] Speake HA, Pereira G, Regan AK. Risk of adverse maternal and foetal outcomes associated with inactivated influenza vaccination in first trimester of pregnancy. Paediatr Perinat Epidemiol. 2021 Mar;35(2):196-205. doi: 10.1111/ppe.12715. Epub 2020 Nov 5. PMID 33155331
- [Background] Idowu MB, Dotters-Katz SK, Kuller JA, Grace MR, Gatta LA. Seasonal Influenza in Pregnancy. Obstet Gynecol Surv. 2025 Jul;80(7):432-442. doi: 10.1097/OGX.0000000000001406. PMID 40598809
- [Background] Wei X, Narasimhan H, Zhu B, Sun J. Host Recovery from Respiratory Viral Infection. Annu Rev Immunol. 2023 Apr 26;41:277-300. doi: 10.1146/annurev-immunol-101921-040450. Epub 2023 Jan 30. PMID 36716750
- [Background] Gandhi L, Maisnam D, Rathore D, Chauhan P, Bonagiri A, Venkataramana M. Respiratory illness virus infections with special emphasis on COVID-19. Eur J Med Res. 2022 Nov 8;27(1):236. doi: 10.1186/s40001-022-00874-x. PMID 36348452
- [Background] Chasekwa B, Munhanzi F, Madhuyu L, Mbewe G, Mabika V, Chidhanguro D, Kofi T, Munengiwa J, Mapfumo H, Musapa M, Shumba S, Hungwe E, Nhokwara M, Bushe N, Kufa R, Mazula P, Chikombingo M, Tengende A, Zanga A, Ziruma A, Bere T, Munyengwa S, Mudimbu C, Murwira Z, Mudzingwa S, Mpofu E, Mutasa B, Sauramba V, Masakadze E, Runodamoto T, Chiorera C, Mushininga A, Bourke CD, Robertson RC, Perussolo J, Donos N, Nyachowe C, Muchekeza M, Chikunya J, Smuk M, Mutasa K, Tavengwa NV, Langhaug LL, Ntozini R, Munjanja SP, Prendergast AJ. A Trial of Trimethoprim-Sulfamethoxazole in Pregnancy to Improve Birth Outcomes. N Engl J Med. 2025 Jun 5;392(21):2125-2134. doi: 10.1056/NEJMoa2408114. PMID 40466066
- [Background] Crump C, Sundquist J, Sundquist K. Adverse Pregnancy Outcomes and Long-Term Mortality in Women. JAMA Intern Med. 2024 Jun 1;184(6):631-640. doi: 10.1001/jamainternmed.2024.0276. PMID 38619848
- [Background] Chen H, Li R, Liu S, Zhao S, Guo T, Tian S, Zhong J, Tang Z, Ge Z, Xia J, Geng T, Pan X, Pan A, Qian F, Liu G. Life's Essential 8 and cardiovascular disease in women with a history of adverse pregnancy outcomes. Eur J Prev Cardiol. 2025 Aug 5;32(10):833-842. doi: 10.1093/eurjpc/zwaf021. PMID 39887026